CLINICAL TRIAL: NCT04680780
Title: Ketogenic Dietary Interventions in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Acronym: Keto-ADPKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Roman Müller, Department II of Internal Medicine, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 02
Record Dates: First submitted 2020-10-01; First posted 2020-12-23 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: ADPKD
Keywords: ADPKD; Ketosis; dietary intervention; ketogenic diet; 3-days water fasting; fasting
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Ketosis; Fasting | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic diet (Experimental): Patients will follow a classical ketogenic diet for 3 month
  Interventions: Other: Ketogenic diet
- 3-days water-fasting (Experimental): Patients will perform water fasting on 3 consecutive days within the first 14 days of each of the 3 months.
  Interventions: Other: 3-days water-fasting
- Control (Placebo Comparator): Patients are allowed to eat ad libitum
  Interventions: Other: Control

INTERVENTIONS:
Other: Ketogenic diet — Patients will follow a classical ketogenic diet for 3 months
  Arms: Ketogenic diet
Other: 3-days water-fasting — Patients will perform water fasting on 3 consecutive days within the first 14 days of each of the 3 months. In one of the 3 months they are - if required - allowed to split the 3 days into periods of 1 and 2 days. On all other days of the intervention period they are allowed to eat ad libitum.
  Arms: 3-days water-fasting
Other: Control — Patients are allowed to eat ad libitum, but will be advised that low salt intake (< 5-7 g/day) and sufficient fluid intake (>3 l/day) which is considered beneficial in ADPKD.
  Arms: Control

SUMMARY:
A mild reduction in food intake significantly inhibits renal cyst growth in mouse models of ADPKD. The underlying mechanism was unknown at the time. Recently published data show that the beneficial effect is not due to caloric restriction per se but due to the induction of the state of ketosis. Dietary interventions leading to ketosis profoundly inhibited renal cyst growth in rodent models of PKD. In addition, acute fasting led to rapid regression of renal cystic burden in mouse, rat and feline models of PKD. Due to these compelling effects in a multitude of PKD animal models, and due to the fact that well-established dietary interventions have a tremendous translational potential, KETO-ADPKD will test such interventions regimens in ADPKD patients.

Two well-established ketogenic dietary regimens will be tested in comparison to a control group to address the following four questions:

1. Feasibility: Are ketogenic dietary interventions acceptable to ADPKD patients in everyday life?
2. Safety: Are there adverse events of ketogenic dietary interventions in ADPKD patients?
3. Efficacy: Do the dietary interventions reach the metabolic endpoints? Do they have a short-term impact on kidney volume?
4. Which of the two diets is the optimal approach?

These questions will be addressed in an exploratory, randomized, open, single center, three-arm dietary intervention study using the following interventions in 21 ADPKD patients per treatment arm:

A) Ketogenic diet B) 3-day water fasting C) Control: ad libitum food intake (no diet)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ADPKD patients (based on genetics or imaging) ≥ 18 and ≤ 60 years
2. Indicators of rapid progression, either of the following:

   * Mayo class 1C-E (measured on screening)
   * Truncating PKD1 mutation,
   * onset of arterial hypertension/urological symptoms < 35 years (patient history)
   * first- or second degree family members reaching ESRD at < 60 years of age (patient history),
   * eGFR loss > 2.5 ml/min/yr (as determined by at least 4 serum creatinine values within the last 4 years, with at least 6 months between each measurement ),
   * PROPKD score > 6 (patient history)
3. CKD-stages G1-3 as determined by eGFR (CKD-EPI)
4. Written informed consent

Exclusion Criteria:

1. Underweight or obese individuals ( as defined by BMI ≤ 18.5 kg/m2 or ≥ 35 kg/m2)
2. Exposure to a ketogenic diet (classical ketogenic diet or modified Atkins)for more than 2 weeks within the last 6 months
3. Participation in a weight-loss program within the last 6 months based on patient history
4. Vegetarian / vegan lifestyle based on patient history
5. Current treatment (or within the last 6 months) with tolvaptan or a somatostatin analogue based on patient history
6. Inability to give informed consent
7. Conditions prohibiting the use of a ketogenic diet (Liver damage, pancreatic failure, pyruvate-carboxylase deficiency, defects in fatty acid oxidation/gluconeogenesis/ketolysis/-neogenesis, hyperinsulinism) based on patient history
8. Diagnosis with any disorder of fatty acid metabolism including Carnitine deficiency (primary), Carnitine palmitoyltransferase (CPT) I or II deficiency, Carnitine translocase deficiency, Beta-oxidation defects, Medium-chain acyl dehydrogenase deficiency (MCAD), Long-chain acyl dehydrogenase deficiency (LCAD), Short-chain acyl dehydrogenase deficiency (SCAD), Long-chain 3-hydroxyacyl-CoA deficiency, Medium-chain 3-hydroxyacyl-CoA deficiency, Pyruvate carboxylase deficiency based on patient history
9. Eating disorder based on patient history (as defined by the assessment of the study physician)
10. Alcohol abuse based on patient history (as defined by the assessment of the study physician)
11. Type 1 diabetes mellitus based on patient history
12. Insulin-dependent type 2 diabetes mellitus based on patient history
13. Contraindication regarding the MRI exam e.g. non-MRI suitable implants ( including cardiac pacemakers, cochlear implants, aneurysm clip), claustrophobia, large tatoos with metal-containing ink
14. Patients, who may be at risk from the blood loss due to scheduled blood draws at the discretion of the physician
15. Pregnancy or breastfeeding
16. Absence of safe contraceptive measures or non-occurrence of menopause (in women)
17. Participation in other interventional trials
18. Persons who are in a dependency/employment relationship with the investigators
19. Accommodation in an institution by judicial or administrative order.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of ketogenic dietary interventions in every-day life, defined as a combination of objective adherence (ketone body levels) and a patient-reported feasibility questionnaire | Day 90
  1. Adherence: (A) Ketogenic diet-group: (1) ketone body levels ≥0.8 mmol/l in ≥75% of blood measurements at visits/patient or (2) ≥10 ppm in ≥75 % of Breathalyzer measurements and ketone body levels ≥0.8 mmol/l in ≥50% of blood measurements at visits/patient, to be reached by ≥ 75% of the participants by ≥50% of all per protocol measurements (B) 3-day water-fasting group:(1) full compliance to diet on ≥75% days/patient (based on diary), to be reached by ≥75% of the participants or by ≥50% of all per protocol measurements (2) at least 1 ketone body level ≥10 ppm/day on at least 2 out of 3 days of each fasting phase (analyzed using breathalyzer).
  2. Patient-reported feasibility will be measured using a dedicated feasibility questionnaire by counting the answers to the questions 1-17 and 21-26 (options ranging from-4 to+4 with higher values indicating better feasibility). Goal: Average value ≥0 in at least 75% of the participants.Both targets have to be met to reach the primary endpoint.

SECONDARY OUTCOMES:
Between group-difference of the relative change in Total kidney volume | baseline and day 90
  Measured by abdominal MRI (segmentation) at screening visit and after the dietary intervention (visit 5).
Between group-difference of the relative change in Body-Mass-Index (BMI) | baseline and day 90
  Determination of BMI before and after dietary intervention
Between group-difference of the relative change of insulin sensitivity | baseline and day 90
  Measurement of insulin-like growth factor (IGF 1), insulin and C-peptide in blood samples (measurement unit µg/l) before and after dietary intervention
Between group-difference in hsCRP | baseline and day 90
  Measurement of high-sensitive CRP (hsCRP) in blood samples before and after dietary intervention
Change in quality of life assessed using the Short Form (12) Health Survey (SF-12) before and after the dietary intervention | Baseline and day 90
  Patients will complete a standardized quality of life questionnaire (QoL, SF-12) before and after the dietary intervention (higher values indicate better QoL, ranging from 0-100)
Change in health-related quality of life assessed using the ADPKD-impact scale before and after the dietary intervention | Baseline and day 90
  Patients will complete a standardized health-related quality of life questionnaire (ADPKD-impact scale) before and after the dietary intervention (lower values indicate better HRQoL, ranging from 1-5)
Between group-difference in blood pressure | Baseline and day 90
  Measurement of systolic and diastolic blood pressure before and after dietary intervention
Incidence of Diet-related Emergent Adverse Events [Safety] at day 30, day 60, day 90 and day 120 | Day 30, day 60, day 90, day 120
  Occurence if Diet-related emergent adverse events will be assessed using lab values (GOT/GPT ≥ 3 times upper limit of normal, increase in serum creatinine fulfilling the KDIGO AKI criteria, triglycerides > 800 mg/dl) and incidence of renal complications (macrohematuria, flank pain, cyst infection, nephrolithiasis)

CONTACTS AND LOCATIONS:
Overall Officials: Roman-Ulrich Müller, Prof., Principal Investigator — Department II of Internal Medicine, University of Cologne
Locations (1):
- Department II of Internal Medicine, University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Cukoski S, Lindemann CH, Arjune S, Todorova P, Brecht T, Kuhn A, Oehm S, Strubl S, Becker I, Kammerer U, Torres JA, Meyer F, Schomig T, Hokamp NG, Siedek F, Gottschalk I, Benzing T, Schmidt J, Antczak P, Weimbs T, Grundmann F, Muller RU. Feasibility and impact of ketogenic dietary interventions in polycystic kidney disease: KETO-ADPKD-a randomized controlled trial. Cell Rep Med. 2023 Nov 21;4(11):101283. doi: 10.1016/j.xcrm.2023.101283. Epub 2023 Nov 7. PMID 37935200